CLINICAL TRIAL: NCT00752752
Title: The Acute Cardiovascular Effects of Marathon Running Using Magnetic Resonance Imaging
Acronym: MARATHON-MRI
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Lihua QU, Coordinator, Corewell Health East
Other Study IDs: HIC2008-083
Record Dates: First submitted 2008-09-12; First posted 2008-09-15 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Myocardial Ischemia; Left Ventricular Systolic Dysfunction; Elevated Cardiac Enzymes
Keywords: Marathon Running; Cardiac Ischemia; Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Ischemia; Ventricular Dysfunction, Left; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Using blood testing and cardiac magnetic resonance imaging (MRI), the investigators aim to determine if there are necrotic areas of myocardium in participants who complete a marathon. In addition, the investigators aim to describe the acute and chronic structural abnormalities that occur as a result of endurance training. The study hypothesis is that myocardial necrosis is present in runners completing a marathon competition.

DETAILED DESCRIPTION:
MARATHON-MI is a prospective, observational study of twenty-five (25) participants with plans of completing the Detroit Free Press Marathon in Detroit, Michigan on October 19, 2008. All participants will undergo a rigorous pre-marathon screening process which will include: 1) blood testing, 2) complete cardiopulmonary exercise testing, 3) ECG testing, 4) Holter monitoring, 5) cardiac MRI. Blood work will be check after the marathon immediately after and one day after the event. Cardiac MRI will be repeated within 12 hours of finishing the marathon. Using the information derived from the blood work and radiological testing, we will attempt to determine if there is an association between marathon running and myocardial necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Detroit Free Press Marathon participant on October 19, 2008,
* Age > 18 years old,
* Ability to provide informed consent.

Exclusion Criteria:

* Known coronary or structural heart disease
* Pregnancy,
* Extreme claustrophobia,
* Metal implants,
* Renal dysfunction.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty-five (25) participants with plans of completing the Detroit Free Press Marathon in Detroit, Michigan on October 19, 2008.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Trivax, MD, Principal Investigator — Physician
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States